CLINICAL TRIAL: NCT00461578
Title: Open Study on the Tolerability and Efficacy of the Combination Chlorproguanil-Dapsone+Artesunate Compared to Amodiaquine+Sulfadoxine-Pyrimethamine for the Treatment of Uncomplicated Falciparum Malaria in Rwandan Children
Brief Title: Tolerability and Efficacy of CD+A Compared to AQ+SP for the Treatment of P.Falciparum Malaria in Rwandan Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDA/RWD/2006
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Malaria
Keywords: P.falciparum; malaria; lapdap+artesunate; safety; efficay
MeSH Terms: conditions — Malaria | interventions — chloroguanil, dapsone drug combination; Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Chlorproguanil-dapsone + artesunate

SUMMARY:
In 2005-2006, a clinical trial was carried out to test safety, tolerability and efficacy of the combination chlorproguanil-dapsone+artesunate (CD+A): 800 children aged 12-59 months with uncomplicated P. falciparum malaria randomly allocated to AQ+SP or CD+A were followed up until day 28 after treatment. Adverse events, clinical and parasitological outcomes were recorded.

DETAILED DESCRIPTION:
Between 2001 and 2006, as an interim strategy, Rwanda chose amodiaquine+ sulfadoxine-pyrimethamine (AQ+SP) as the first line anti-malaria treatment. Although the clinical response to this combination was relatively good in 2001, since then its efficacy has steadily declined: in 2002 the proportion of successful treatment (recorded at 28 days and PCR-unadjusted) was 83 % (Rwagacondo et al., 2003) and in 2003 it was 74% (Karema et al., 2006). Different artemisinin-based combination treatments (ACTs) such as amodiaquine+artesunate (AQ+AS), dihydroartemisinin-piperaquine (DHAPPQ) and artemether-lumefantrine (ALN) have been tested in the past few years as possible alternatives to AQ+SP (Fanello et al., 2006; Karema et al., 2006).

Chlorproguanil-dapsone (also known asLapDap) is an antifolate combination similar to sulfadoxine/pyrimethamine (SP) but for two important features: (1) it is rapidly eliminated and therefore exerts less selective pressure for resistance-conferring parasite mutations than does SP (Winstanley et al., 1997; Nzila et al., 2000b) and (2) it is active against the SP-resistant forms of the parasite that are found in Africa (Mutabingwa et al., 2001a,b; Kublin et al., 2002). Moreover, a pediatric course of treatment of LapDap is estimated to cost $0.15 (Mutabingwa et al., 2001b), making it orders of magnitude less expensive than any marketed antimalarial drug other than chloroquine and SP.

In 2005-2006, a clinical trial was carried out to test safety, tolerability and efficacy of the combination chlorproguanil-dapsone+artesunate (CD+A): 800 children aged 12-59 months with uncomplicated P. falciparum malaria randomly allocated to AQ+SP or CD+A were followed up until day 28 after treatment. Adverse events, clinical and parasitological outcomes were recorded.

Based on the results of all trials carried out by the NMCP, The Rwandan Ministry of Health has now changed the first line to artemether-lumefantrine (ALN), Coartem®. The drug arrived in the country in October 2006.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-59 months;
* Weight ≥5 kg;
* Monoinfection with P. falciparum;
* Parasite density between 2,000-200,000/µL;
* Fever (axillary body temperature =>37.5C) or history of fever in the preceding 24 hours;
* Packed Cell Volume (PCV) >21%.

Exclusion Criteria:

* Severe malaria;
* Mixed malaria infection;
* Any other concomitant illness or underlying disease;
* Known allergy to the study drugs being used in this trial;
* Clear history of adequate antimalarial treatment in the previous 72 hours.

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800
Dates: Start 2005-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Incidence of microscopically and genotypically confirmed recrudescent infections in the different treatment groups by day 28

SECONDARY OUTCOMES:
Parasite clearance
Fever clearance
Occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Umberto d'Alessandro, MD, Study Director — ITM
Locations (1):
- Programme Nationale Integre de Lutte contre le Paludisme, Kigali, Rwanda

REFERENCES:
- [Derived] Fanello CI, Karema C, Avellino P, Bancone G, Uwimana A, Lee SJ, d'Alessandro U, Modiano D. High risk of severe anaemia after chlorproguanil-dapsone+artesunate antimalarial treatment in patients with G6PD (A-) deficiency. PLoS One. 2008;3(12):e4031. doi: 10.1371/journal.pone.0004031. Epub 2008 Dec 29. PMID 19112496
- [Derived] Fanello CI, Karema C, Ngamije D, Uwimana A, Ndahindwa V, Van Overmeir C, Van Doren W, Curtis J, D'Alessandro U. A randomised trial to assess the efficacy and safety of chlorproguanil/dapsone + artesunate for the treatment of uncomplicated Plasmodium falciparum malaria. Trans R Soc Trop Med Hyg. 2008 May;102(5):412-20. doi: 10.1016/j.trstmh.2008.01.013. Epub 2008 Mar 6. PMID 18328518